CLINICAL TRIAL: NCT00572689
Title: Pilot Study of Exenatide Pharmacokinetics and Pharmacodynamics in Gestational Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Jason Umans, Prinipal Investigator, Georgetown University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Exenatide.GDM; 202-801-2636
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Gestational Diabetes
Keywords: Exenatide; TCF7L2 polymorphism; Pharmacodynamics; Pharmacokinetics
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Subject receives injection of 10 micrograms of Exenatide sub-cutaneously the given mixed meal test and blood samples will be drawn for laboratory testing.
  Interventions: Drug: Exenatide; Genetic: Buccal/blood Sample Collection
- B (No Intervention): Patients given mixed meal test and blood samples drawn for laboratory testing

INTERVENTIONS:
Drug: Exenatide — 10 microgram injected sub-cutaneously once
  Other Names: Byetta
  Arms: A
Genetic: Buccal/blood Sample Collection — Buccal/blood Sample collection for TCF7L2 polymorphism genetic testing
  Arms: A

SUMMARY:
This study is being done to study how exenatide, an FDA-approved drug that lowers blood sugar in non-pregnant patients with type II diabetes, works in pregnant women. To do this, we will study the drug's pharmacokinetics (what the body does to the drug; specifically, how quickly your body breaks down and excretes exenatide) and pharmacodynamics (what the drug does to the body; specifically, how effectively exenatide helps your pancreas secrete insulin and how well it controls blood sugar after a meal). There are only two main drug therapies (insulin injections and glyburide pills) currently used for gestational diabetes and not all women achieve good enough blood sugar control without side effects. Therefore, we hope to find out if exenatide might also be helpful in gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (singleton)
* Gestational diabetes not requiring medical therapy
* Between 18 and 50 years of age
* Able to give written informed consent

Exclusion Criteria:

* Women in the first trimester of pregnancy
* Hematocrit less than 30%
* Current or past treatment with any hypoglycemic agent
* Women with gastrointestinal disease or symptoms consistent with nausea, vomiting, abdominal pain or reflux requiring medical treatment.
* Women with high triglyceride levels, history of gallbladder or pancreatic disease.
* Clinical diagnosis or history of any renal insufficiency (or decreased creatinine clearance)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
glycemic control through insulin, glucose, c-peptide and glucagon assays | duing testing days

SECONDARY OUTCOMES:
TCF7L2 polymorphism | During subject testing days
Exenatide Pharmacodynamics and Pharmacokinetics | During testing days

CONTACTS AND LOCATIONS:
Overall Officials: Jason G Umans, MD, PhD, Principal Investigator — Georgetown University Medical Center, Medstar Health Research Institute; Maisa N Feghali, MD, Study Director — Medstar Health Research Institute
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia